CLINICAL TRIAL: NCT05986669
Title: Safety and Effectiveness of DSP Dental Implant Systems: Prospective Study Multicenter Involving Real-world Data
Status: Recruiting | Type: Observational
Sponsor: DSP Industrial Ltda (Industry)
Responsible Party: Sponsor
Other Study IDs: DSP_001
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-08

CONDITIONS: Dental Implant
Keywords: Dental Implants; Dental Prostheses; Safety and efficacy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Studies on facial trauma are essential to establish an appropriate treatment approach, assess the ability to restore functions and seek ways of prevention. Among craniofacial injuries, fractures of the zygomatic complex are the most frequent, occurring in 25-30% of cases. Statistical analysis shows that traffic collisions (41%), domestic accidents (23%) and sports accidents (18%) are the main causes. Dental implants have emerged as a rehabilitative alternative for these patients, being considered the first choice for individuals who have lost all or part of their dental arch. In addition to providing a better quality of life, it reconstitutes masticatory function, self-esteem and phonetics. Understanding the importance of evaluating the performance of dental implants and considering the responsibility for the health of patients, there was a need to evaluate the effectiveness and safety of the Standard Internal Hexagon Implant System (HIS), Large Internal Hexagon (HIL), Flexcone (FC) , Mini Flexcone (FCM) and Morse Internal Hexagon, from DSP. In this prospective study, 1053 implants will be included. To be eligible, patients can be of both sexes, be 18 years of age or older, any race and gender, have partial or total tooth loss, present good local and general health conditions and psychological disposition to undergo common oral surgery procedures. under local anesthesia and healthy edentulous region as they will be subsequently submitted to surgical procedures using the DSP Implant System. Electronic data collection and management will be performed using the REDCap software, with categorical variables being described as absolute and relative frequencies and continuous ones being tested for normality using the Shapiro-Wilk test. Osseointegration percentages between 30 days and 6 months will also be calculated. Other efficacy outcomes and incidence of adverse events will be estimated with 95% confidence intervals. As a result, from the strengthening of product evaluation actions, it is expected to demonstrate that the implant has a good safety and efficacy profile to be offered to the population.

DETAILED DESCRIPTION:
The study was designed as a prospective observational clinical record. This protocol will be submitted to the Ethics Committee and patients will be included only after ethics committee approval. All data will be collected from procedures performed in actual clinical practice. Specific surgical interventions will not be performed for the purposes of this study, since this is an observational study.

After the surgeries, the patients will be followed up for one year. The patient's data will be collected on five visits scheduled for assessment of the outcomes of the study. (Baseline, T0, T90, T180 and T360).

The forecast for the study end is 24 months after the first inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes will be included;
* Regardless of race/color;
* Aged between 18 and 70 years;
* Who present partial or total tooth loss in a minimum period of three months;
* Healthy edentulous region;
* Good local and general health conditions, and psychological disposition;
* To undergo common oral surgery procedures, under local anesthesia, in addition to undergoing surgical procedures using one of the implant systems under evaluation (Standard Internal Hexagon (HIS); Large Internal Hexagon (HIL); Flexcone (FC); Flexcone Mini (FCM) and Morse Internal Hexagon (HIM).

Exclusion Criteria:

* Patients who need bone grafting;
* Smokers who smoke 10 cigarettes/day or more;
* Individuals who make continuous use of bisphosphonates and anticoagulants, alcoholics, and/or users of illicit drugs
* Pregnant women;
* Diabetics with uncontrolled glycemia and individuals
* Patientes who were treated with radiotherapy.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients to study will be recruited from the site UNESP and DSP Training Center according to the inclusion and exclusion criteria shown in the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Implant success rate 6 months after the procedure | 6 months
  Success = no radiolucency, no mobility, no recurrent peri-implant infection, no persistent pain

SECONDARY OUTCOMES:
Adverse events related to medical device or procedure | Through study completion, an average of 2 years
  Record of events that may happen

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo C Goiato, PhD, Principal Investigator — UPECLIN HC FM Botucatu Unesp; Rafael Correira, PhD, Principal Investigator — DSP
Locations (2):
- Brazil (2):
  - DSP Oral Clinica, Campo Largo, Paraná
  - Universidade Estadual Paulista (UNESP), São Paulo, São Paulo